CLINICAL TRIAL: NCT01582945
Title: N-methyl-D-aspartate Antagonist (Ketamine) Infusion for Treatment-resistant Major Depressive Disorder With Suicidal Ideation
Brief Title: Ketamine Infusion for Treatment-resistant Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Instructor HMS, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-002800
Record Dates: First submitted 2012-04-17; First posted 2012-04-23 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: Treatment resistant; suicidal ideation; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine IV (Experimental): Patients will receive open label augmentation with IV Ketamine at 0.5mg/kg, twice a week for 3 weeks
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine IV 0.5mg/kg infusion twice a week for 3 weeks as augmentation of ongoing antidepressant regimen

SUMMARY:
Ketamine infusion has been shown to have rapid antidepressant properties, however the possible use of ketamine in treatment-resistant depression as augmentation has not been investigated. The overall aim of this study is to assess the feasibility, safety and tolerability, efficacy and duration of the effect of intravenous N-methyl-D-aspartate antagonist ketamine as augmentation of antidepressants for chronic suicidal ideation in subjects with severe treatment-resistant depression (TRD).

This is an open-label study (pilot).

DETAILED DESCRIPTION:
Patients will undergo two weeks of prospective observation, they will then receive ketamine IV 0.5mg/kg over 45 minutes as augmentation of their ongoing antidepressant regimen; after three infusions this dose will be increased increase to 0.75 mg/kg in non-responders. The schedule of administration will be twice a week for 3 weeks. After this phase, the patient will be followed with assessments every two weeks for three months.

Total duration of the study is 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with severe treatment-resistant MDD
* Currently depressed
* Currently under regular psychiatric care
* On an aggressive antidepressant regimen, stable for 4 weeks

Exclusion Criteria:

* No history of other major psychiatric illnesses, including bipolar disorder
* No history of psychosis
* No history of drug abuse
* No major medical illness or unstable medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, MD, Principal Investigator — MGH Department of Psychiatry
Locations (1):
- Depression Clinical and Research Program - MGH, Boston, Massachusetts, United States

REFERENCES:
- [Result] Ionescu DF, Swee MB, Pavone KJ, Taylor N, Akeju O, Baer L, Nyer M, Cassano P, Mischoulon D, Alpert JE, Brown EN, Nock MK, Fava M, Cusin C. Rapid and Sustained Reductions in Current Suicidal Ideation Following Repeated Doses of Intravenous Ketamine: Secondary Analysis of an Open-Label Study. J Clin Psychiatry. 2016 Jun;77(6):e719-25. doi: 10.4088/JCP.15m10056. PMID 27232360
- [Result] Cusin C, Ionescu DF, Pavone KJ, Akeju O, Cassano P, Taylor N, Eikermann M, Durham K, Swee MB, Chang T, Dording C, Soskin D, Kelley J, Mischoulon D, Brown EN, Fava M. Ketamine augmentation for outpatients with treatment-resistant depression: Preliminary evidence for two-step intravenous dose escalation. Aust N Z J Psychiatry. 2017 Jan;51(1):55-64. doi: 10.1177/0004867416631828. PMID 26893373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were referred to the study by their primary psychiatrists and no compensation was provided for participation.
Pre-assignment Details: Subjects underwent a psychiatric screening evaluation, physical exam, EKG, laboratory testing, and a urine screening for substances of abuse to determine study eligibility.
Groups:
- Treatment-resistant Depression Patients: Outpatient sample of patients (18-65 years old) with treatment-resistant major depressive disorder (TRD).
Period: Overall Study
Arm/Group | Treatment-resistant Depression Patients
Started | 14
Completed | 12
Not Completed | 2
Not completed — Intolerable side-effects | 1
Not completed — Scheduling conflicts | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment-resistant Depression Patients
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 14
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — Scores may range from 0-81 with higher scores indicate greater depression severity. In order to be included in the study, participants must have had a Hamilton Depression Rating Scale-28 items (HAM-D28) score ⩾20 at screening.
  units on a scale | 28.6 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Response to Ketamine as Measured by Hamilton Depression Rating Scale -28 Items (HAMD28)
Description: Patients will be assessed with HAMD-28 weekly for the first 8 weeks, then every two weeks for another 8 weeks. Participants were considered as responders if there was a ⩾50% improvement on the HAM-D28.
Time Frame: Weekly for total duration of 4 months
Population: The subjects received a total of 6 infusions, twice a week for three weeks.
Measure: Number; unit: participants who met response criteria
Groups:
- Ketamine IV: Patients will receive open label augmentation with IV Ketamine at 0.5mg/kg over the course of 45 minutes, twice a week for 3 weeks. Participants received this dosage for the first three of six IV ketamine infusions. If participants do not experience an improvement of greater or equal to 30% in HAM-D scores after the first three infusions, the dose will be increased to 0.75mg/kg for the subsequent three infusions.
  Ketamine: Ketamine IV 0.5mg/kg infusion twice a week for 3 weeks as augmentation of ongoing antidepressant regimen
Arm/Group | Ketamine IV
Number analyzed (Participants) | 12
participants who met response criteria | 5

ADVERSE EVENTS:
Arm/Group | Ketamine IV
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No